CLINICAL TRIAL: NCT05603819
Title: Clinical Validation Study for EDIT-B Test: an Aid for Differential Diagnosis of Bipolar Disorder, Based on RNA Editing Blood Biomarkers
Acronym: EDIT-B
Status: Completed | Type: Observational
Sponsor: Alcediag (Industry)
Collaborators: Hospital Clinic of Barcelona (Other); Fundacion Clinic per a la Recerca Biomédica (Other); Region Capital Denmark (Other); GHU Paris Psychiatry & Neurosciences (Other); Parc Sanitari Sant Joan de Déu (Other); Fundació Sant Joan de Déu (Other); Synlab Italie (Unknown)
Responsible Party: Sponsor
Other Study IDs: EDIT-B
Record Dates: First submitted 2022-10-28; First posted 2022-11-03 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Bipolar Disorder; Major Depressive Disorder
MeSH Terms: conditions — Bipolar Disorder; Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood samples (2x0.5 mL) stored in PAXgene RNA collection tubes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bipolar disorder: Patients with depression suffering from bipolar disorder.
  Interventions: Device: EDIT-B
- Major depressive disorder: Patients with depression suffering from major depressive disorder.
  Interventions: Device: EDIT-B

INTERVENTIONS:
Device: EDIT-B — To perform EDIT-B test, questionnaires and 2x0.5 mL whole blood are collected from each patient.

SUMMARY:
Differentiation between major depressive disorder (MDD) and bipolar disorder (BD) as soon as possible in the patient journey represents a major clinical issue. When the patient is in a depressive phase, the symptoms are similar between the two pathologies and the current clinical scales fail in distinguishing them. Physicians often report this difficulty and as a consequence, the mean time from onset to bipolar disorder diagnosis is currently 7.5 years. These diagnostic delays and misdiagnosis lead to damaging consequences for patients and their loved ones: worsening of symptoms, comorbidities, suicide risk and inadequate care resulting in severe impairment in social and occupational functioning. Faced with these high expectations for accurate diagnostic methods for an earlier management of psychiatric patients, the combination of relevant clinical features and biomarkers could stand for a solution, leading to a personalised approach in patients with mood disorders.

In a first clinical discovery study, a panel of RNA biomarkers in the blood of patients with a major depressive episode (MDE) has been identified, allowing to differentiate bipolar disorder from MDD (unipolar depression). These biomarkers are based on RNA modifications, namely RNA editing, that could be identified using molecular biology, NGS and artificial intelligence. This panel constitutes EDIT-B test, which is based on Alcediag's proprietary and patented biomarkers and algorithms.

The present study aims to validate the biomarker signatures proposed by Alcediag by measuring the association between the modifications of the RNA editing and major depressive disorder/ bipolar disorder diagnosis, in patients with a MDE in real-life setting pilot centres.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Male or female ≥ 18 and ≤ 80 years of age at inclusion.
3. MADRS ≥ 20
4. In- and out-patients can be recruited.
5. Diagnosed with MDE with the MINI for DSM-5
6. Currently treated for the MDE
7. Diagnosed with MDD or BD with the MINI for DSM-5.
8. For patients with BD: at least one manic or hypomanic episode
9. For patients with MDD: at least one MDE

Exclusion Criteria:

1. MDD patients with first degree family history of bipolar disorder
2. YMRS > 12
3. Pregnant women
4. Unipolar or bipolar depression secondary to major central nervous system affections, including infections in the brain, tumours of the brain, stroke, Alzheimer's disease, Parkinson's disease, Multiple sclerosis, other major brain affections
5. Schizo-affective patients

Abbrevations:

BD Bipolar Disorder DSM-5 Diagnostic and Statistical Manual of Mental disorders 5 MADRS Montgomery-Asberg Depression Rating Scale MDD Major Depressive Disorder MDE Major Depressive Episode MINI Mini-International Neuropsychiatric Interview YMRS Young Mania Rating Scale

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with depression meeting the MDE criteria in DSM-5 using the MINI will be eligible for the study. They can be in- and out-patients for each clinical center.
Sampling Method: Probability Sample
Enrollment: 418 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Diagnostic performances of EDIT-B signatures on MDD vs. BD differentiation in patients with depression. | Specimen collection needed for evaluation of diagnostic performances: 1 day (= 1 visit).
  The objective of this study is to estimate three EDIT-B signatures in term of their external validity. For this purpose, performances of the tests will be estimated by calculating for each signature its Sensitivity (i.e. the probability that a test will indicate 'bipolar disorders' among those with this disease), Specificity (i.e. the fraction of those without bipolar disorders who will have a negative test result) and its Accuracy to predict the diagnosis of bipolar disorders. In addition, Area under the ROC curves of each EDIT-B signature will be calculated.
  The categorisation of the type of disorder (MDD vs. BD) by experts will be based on the MINI considered as the gold standard for diagnosis.
  The performances of the tested signatures will be compared on a two-by-two basis by comparing sensitivities and specificity , using the methods based on Mac Nemar test proposed by Hawass. AUC-ROC of the 3 signatures will also be compared by DeLong method.

CONTACTS AND LOCATIONS:
Overall Officials: Eduard Vieta, Principal Investigator — Hospital Clinic of Barcelona
Locations (4):
- The Capital Region of Denmark, Copenhagen, Denmark
- GHU Paris Psychiatrie & Neurosciences, Paris, France
- Spain (2):
  - Parc Sanitari Sant Joan de Déu, Sant Boi de Llobregat, Barcelona
  - Hospital Clínic de Barcelona, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salvetat N, Checa-Robles FJ, Patel V, Cayzac C, Dubuc B, Chimienti F, Abraham JD, Dupre P, Vetter D, Mereuze S, Lang JP, Kupfer DJ, Courtet P, Weissmann D. A game changer for bipolar disorder diagnosis using RNA editing-based biomarkers. Transl Psychiatry. 2022 May 4;12(1):182. doi: 10.1038/s41398-022-01938-6. PMID 35504874
- [Background] Montgomery SA, Asberg M. A new depression scale designed to be sensitive to change. Br J Psychiatry. 1979 Apr;134:382-9. doi: 10.1192/bjp.134.4.382. PMID 444788
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Young RC, Biggs JT, Ziegler VE, Meyer DA. A rating scale for mania: reliability, validity and sensitivity. Br J Psychiatry. 1978 Nov;133:429-35. doi: 10.1192/bjp.133.5.429. PMID 728692
- [Background] Kim SH, Kim HJ, Lee SI, Jo MW. Comparing the psychometric properties of the EQ-5D-3L and EQ-5D-5L in cancer patients in Korea. Qual Life Res. 2012 Aug;21(6):1065-73. doi: 10.1007/s11136-011-0018-1. Epub 2011 Sep 23. PMID 21947656
- [Background] Hawass NE. Comparing the sensitivities and specificities of two diagnostic procedures performed on the same group of patients. Br J Radiol. 1997 Apr;70(832):360-6. doi: 10.1259/bjr.70.832.9166071.
- [Background] DeLong ER, DeLong DM, Clarke-Pearson DL. Comparing the areas under two or more correlated receiver operating characteristic curves: a nonparametric approach. Biometrics. 1988 Sep;44(3):837-45. PMID 3203132
- [Background] Buderer NM. Statistical methodology: I. Incorporating the prevalence of disease into the sample size calculation for sensitivity and specificity. Acad Emerg Med. 1996 Sep;3(9):895-900. doi: 10.1111/j.1553-2712.1996.tb03538.x. PMID 8870764
- [Background] Merikangas KR, Jin R, He JP, Kessler RC, Lee S, Sampson NA, Viana MC, Andrade LH, Hu C, Karam EG, Ladea M, Medina-Mora ME, Ono Y, Posada-Villa J, Sagar R, Wells JE, Zarkov Z. Prevalence and correlates of bipolar spectrum disorder in the world mental health survey initiative. Arch Gen Psychiatry. 2011 Mar;68(3):241-51. doi: 10.1001/archgenpsychiatry.2011.12. PMID 21383262
- [Background] Carvalho AF, Solmi M, Sanches M, Machado MO, Stubbs B, Ajnakina O, Sherman C, Sun YR, Liu CS, Brunoni AR, Pigato G, Fernandes BS, Bortolato B, Husain MI, Dragioti E, Firth J, Cosco TD, Maes M, Berk M, Lanctot KL, Vieta E, Pizzagalli DA, Smith L, Fusar-Poli P, Kurdyak PA, Fornaro M, Rehm J, Herrmann N. Evidence-based umbrella review of 162 peripheral biomarkers for major mental disorders. Transl Psychiatry. 2020 May 18;10(1):152. doi: 10.1038/s41398-020-0835-5. PMID 32424116
- [Background] Carvalho AF, Firth J, Vieta E. Bipolar Disorder. N Engl J Med. 2020 Jul 2;383(1):58-66. doi: 10.1056/NEJMra1906193. No abstract available. PMID 32609982
- [Background] Fiedorowicz JG, He J, Merikangas KR. The association between mood and anxiety disorders with vascular diseases and risk factors in a nationally representative sample. J Psychosom Res. 2011 Feb;70(2):145-54. doi: 10.1016/j.jpsychores.2010.07.010. Epub 2010 Sep 18. PMID 21262417
- [Background] Pan JX, Xia JJ, Deng FL, Liang WW, Wu J, Yin BM, Dong MX, Chen JJ, Ye F, Wang HY, Zheng P, Xie P. Diagnosis of major depressive disorder based on changes in multiple plasma neurotransmitters: a targeted metabolomics study. Transl Psychiatry. 2018 Jul 10;8(1):130. doi: 10.1038/s41398-018-0183-x. PMID 29991685
- [Background] Kessing LV. Course and cognitive outcome in major affective disorder. Dan Med J. 2015 Nov;62(11):B5160. PMID 26522485
- [Background] Giridharan VV, Sayana P, Pinjari OF, Ahmad N, da Rosa MI, Quevedo J, Barichello T. Postmortem evidence of brain inflammatory markers in bipolar disorder: a systematic review. Mol Psychiatry. 2020 Jan;25(1):94-113. doi: 10.1038/s41380-019-0448-7. Epub 2019 Jun 27. PMID 31249382
- [Background] Maes M, Carvalho AF. The Compensatory Immune-Regulatory Reflex System (CIRS) in Depression and Bipolar Disorder. Mol Neurobiol. 2018 Dec;55(12):8885-8903. doi: 10.1007/s12035-018-1016-x. Epub 2018 Apr 2. PMID 29611101
- [Background] Mannion NM, Greenwood SM, Young R, Cox S, Brindle J, Read D, Nellaker C, Vesely C, Ponting CP, McLaughlin PJ, Jantsch MF, Dorin J, Adams IR, Scadden AD, Ohman M, Keegan LP, O'Connell MA. The RNA-editing enzyme ADAR1 controls innate immune responses to RNA. Cell Rep. 2014 Nov 20;9(4):1482-94. doi: 10.1016/j.celrep.2014.10.041. Epub 2014 Nov 13. PMID 25456137
- [Background] Lamers MM, van den Hoogen BG, Haagmans BL. ADAR1: "Editor-in-Chief" of Cytoplasmic Innate Immunity. Front Immunol. 2019 Jul 25;10:1763. doi: 10.3389/fimmu.2019.01763. eCollection 2019. PMID 31404141
- [Background] Rosenthal JJ, Seeburg PH. A-to-I RNA editing: effects on proteins key to neural excitability. Neuron. 2012 May 10;74(3):432-9. doi: 10.1016/j.neuron.2012.04.010. PMID 22578495
- [Background] Berg KA, Cropper JD, Niswender CM, Sanders-Bush E, Emeson RB, Clarke WP. RNA-editing of the 5-HT(2C) receptor alters agonist-receptor-effector coupling specificity. Br J Pharmacol. 2001 Sep;134(2):386-92. doi: 10.1038/sj.bjp.0704255. PMID 11564657
- [Background] Yang W, Wang Q, Kanes SJ, Murray JM, Nishikura K. Altered RNA editing of serotonin 5-HT2C receptor induced by interferon: implications for depression associated with cytokine therapy. Brain Res Mol Brain Res. 2004 Apr 29;124(1):70-8. doi: 10.1016/j.molbrainres.2004.02.010. PMID 15093687
- [Background] Chimienti F, Cavarec L, Vincent L, Salvetat N, Arango V, Underwood MD, Mann JJ, Pujol JF, Weissmann D. Brain region-specific alterations of RNA editing in PDE8A mRNA in suicide decedents. Transl Psychiatry. 2019 Feb 15;9(1):91. doi: 10.1038/s41398-018-0331-3. PMID 30770787
- [Background] Weissmann D, van der Laan S, Underwood MD, Salvetat N, Cavarec L, Vincent L, Molina F, Mann JJ, Arango V, Pujol JF. Region-specific alterations of A-to-I RNA editing of serotonin 2c receptor in the cortex of suicides with major depression. Transl Psychiatry. 2016 Aug 30;6(8):e878. doi: 10.1038/tp.2016.121. PMID 27576167
- [Background] Bender AT, Beavo JA. Cyclic nucleotide phosphodiesterases: molecular regulation to clinical use. Pharmacol Rev. 2006 Sep;58(3):488-520. doi: 10.1124/pr.58.3.5. PMID 16968949
- [Background] Salvetat N, Van der Laan S, Vire B, Chimienti F, Cleophax S, Bronowicki JP, Doffoel M, Bourliere M, Schwan R, Lang JP, Pujol JF, Weissmann D. RNA editing blood biomarkers for predicting mood alterations in HCV patients. J Neurovirol. 2019 Dec;25(6):825-836. doi: 10.1007/s13365-019-00772-9. Epub 2019 Jul 22. PMID 31332697
- [Background] Salvetat N, Chimienti F, Cayzac C, Dubuc B, Checa-Robles F, Dupre P, Mereuze S, Patel V, Genty C, Lang JP, Pujol JF, Courtet P, Weissmann D. Phosphodiesterase 8A to discriminate in blood samples depressed patients and suicide attempters from healthy controls based on A-to-I RNA editing modifications. Transl Psychiatry. 2021 Apr 30;11(1):255. doi: 10.1038/s41398-021-01377-9. PMID 33931591
- [Background] Wang P, Yu S, Liu J, Zhang D, Kang X. Seven novel mutations of ADAR in multi-ethnic pedigrees with dyschromatosis symmetrica hereditaria in China. Mol Genet Genomic Med. 2019 Oct;7(10):e00905. doi: 10.1002/mgg3.905. Epub 2019 Aug 18. PMID 31423758
- [Background] Jones SR, Carley S, Harrison M. An introduction to power and sample size estimation. Emerg Med J. 2003 Sep;20(5):453-8. doi: 10.1136/emj.20.5.453. PMID 12954688
- [Derived] Miranda-Mendizabal A, Vetter D, Zambrano J, Zarp J, Chavarria V, Gimenez-Palomo A, Gonzalez-Campos M, Valenti M, Walczer Baldinazzo L, Siddi S, Ferrari M, Weissmann D, Henry C, Haro JM, Vedel Kessing L, Vieta E. RNA editing-based biomarker blood test for the diagnosis of bipolar disorder: protocol of the EDIT-B study. Ann Gen Psychiatry. 2025 Feb 6;24(1):7. doi: 10.1186/s12991-024-00544-8. PMID 39915772